CLINICAL TRIAL: NCT02644967
Title: A Phase 1/2 Study to Assess the Safety and Efficacy of Intratumoral IMO-2125 in Combination With Ipilimumab or Pembrolizumab in Patients With Metastatic Melanoma (ILLUMINATE-204)
Brief Title: A Phase 2 Study to Assess the Safety and Efficacy of IMO-2125 With 8 mg Ipilimumab in Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Idera Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2125-204; ILLUMINATE-204 (Other: Idera Pharmaceuticals, Inc.)
Record Dates: First submitted 2015-12-23; First posted 2016-01-01 (Estimated); Results first posted 2022-08-03 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-07

CONDITIONS: Metastatic Melanoma
Keywords: ILLUMINATE- 204; IMO-2125; tilsotolimod
MeSH Terms: conditions — Melanoma | interventions — tilsotolimod; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Phase 2, 8 mg Tilso/Ipi (Experimental): IMO-2125 intratumoral injection plus ipilimumab
  Interventions: Drug: IMO-2125; Drug: Ipilimumab

INTERVENTIONS:
Drug: IMO-2125 — Drug: IMO-2125 Intratumoral injection administered as 9 doses on Weeks 1, 2, 3, 5, 8, 11, 17, 23, and 29.
  Other Names: tilsotolimod (tilso)
Drug: Ipilimumab — 4 doses administered intravenously at a dose of 3 mg/kg over 90 minutes on Weeks 2, 5, 8, and 11.
  Other Names: Yervoy®

SUMMARY:
The goal of the Phase 1 study was to find the recommended Phase 2 dose of the study drug IMO-2125 (tilsotolimod) that can be given in combination with ipilimumab (ipi) or pembrolizumab (pembro) to participants with metastatic melanoma and assess the safety, tolerability, pharmacokinetics (PK), and immunogenicity when administered in combination with ipilimumab or pembrolizumab.

DETAILED DESCRIPTION:
The open-label single-arm Phase 2 study was designed to assess the recommended dose for safety, tolerability, pharmacokinetics (PK), immunogenicity, and efficacy of 8 mg IMO-2125 (tilsotolimod) when administered in combination with ipilimumab.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically confirmed metastatic melanoma with measurable, stage III (lymph node or in transit lesions) or stage IVA, IVB, or IVC disease.
2. Patients must have symptomatic or radiographic progression during or after treatment with a PD-(L)1 inhibitor administered either as monotherapy or in combination.

   1. The interval between last PD-(L)1 directed treatment and start of study treatment should be at least 21 days.
   2. Prior BRAF or MEK inhibitor treatment is not required. However, for patients with known BRAF status:

      * Those with BRAF wild type may have had a maximum of two previous systemic regimens for the treatment of melanoma.
      * Those with a BRAF mutation may have had a maximum of three previous systemic regimens for the treatment of melanoma.
   3. Prior ipilimumab is permitted.
   4. Previous treatment with either a PD-1 inhibitor (for patients enrolling on the IMO-2125 + pembrolizumab combination) or CTLA-4 inhibitor (for patients enrolling on the IMO-2125 + ipilimumab combination if applicable) should not have been accompanied by DLT for which permanent discontinuation is recommended (per USPI).

      * Patients with a history of Grade ≥2 gastrointestinal symptoms (e.g., diarrhea, colitis) during prior checkpoint inhibitor treatment should be discussed with the Idera Medical Monitor during the Screening Period before starting study treatment.
3. Phase 1 patients must have at least two measurable tumor lesions ≥ 1.0 cm that are accessible to biopsy. Phase 2 patients must have at least one measurable lesion (per RECIST v1.1) which may be the same site that is used for the intratumoral injections.
4. Patients must be ≥ 18 years of age.
5. Patients must have Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2.
6. Patients must meet the following laboratory criteria:

   1. Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L (1500/mm3)
   2. Platelet count ≥ 75 x 10^9/L (75,000/mm3)
   3. Hemoglobin ≥ 8.0 g/dL (4.96 mmol/L)
   4. Serum creatinine ≤ 1.5 x upper limit of normal (ULN) or calculated creatinine clearance ≥ 60 mL/minute
   5. Aspartate aminotransferase (AST) ≤ 2.5 x ULN; alanine aminotransferase (ALT) ≤ 2.5 x ULN; AST/ALT < 5 x ULN if liver involvement
   6. Serum bilirubin ≤ 1.5 x ULN, except in patients with Gilbert's Syndrome who must have a total bilirubin < 3 mg/dL
7. Women of childbearing potential (WOCBP) and men must agree to use effective contraceptive methods from Screening throughout the study treatment period and until at least 90 days after the last dose of IMO-2125, 3 months after the last dose of ipilimumab or at least 4 months after the last dose of pembrolizumab.
8. Patients must have an anticipated life expectancy > 3 months.

Exclusion Criteria:

1. Patients who have received prior therapy with a TLR agonist, excluding topical agents. Patients who have received experimental vaccines or other investigational immune therapies should be discussed with the Medical Monitor to confirm eligibility.
2. Patients who have received systemic treatment with IFN-α within the previous 6 months prior to enrolling into this study.
3. Patients with known hypersensitivity to any oligodeoxynucleotide.
4. Patients with active autoimmune disease requiring disease-modifying therapy.
5. Patients requiring concurrent systemic steroid therapy higher than physiologic dose (7.5 mg/day of prednisone).
6. Patients with any form of active primary or secondary immunodeficiency.
7. Patients with another primary malignancy that has not been in remission for at least 3 years.
8. Patients with active systemic infections requiring antibiotics or active hepatitis A, B, or C.
9. Patients with a known diagnosis of human immunodeficiency virus (HIV) infection.
10. Patients who previously had a severe reaction to treatment with a human antibody.
11. Patients with known central nervous system, meningeal, or epidural disease.
12. Women who are pregnant or breastfeeding.
13. Patients with impaired cardiac function or clinically significant cardiac disease.
14. Patients with ocular melanoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2020-02 (Actual); Study Completion 2021-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Idera Medical Director, Study Director — Idera Pharmaceuticals, Inc.
Locations (10):
- United States (10):
  - The University of Arizona Cancer Center, Tucson, Arizona
  - Moffitt Cancer Center Research Institute, Tampa, Florida
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Cancer Center, Westwood, Kansas
  - Roswell Park Cancer Institute, Buffalo, New York
  - Icahn School Of Medicine at Mount Sinai, New York, New York
  - Gabrail Cancer Center, Canton, Ohio
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - University of Utah- Huntsman Cancer Institute, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The Phase 2 study was conducted at nine (9) academic cancer centers.
Pre-assignment Details: In the Phase 2 study, all participants were assigned to a single arm and received IMO-2125 (tilsotolimod [tilso]) at the recommended Phase 2 dose (RP2D) of 8 mg, in combination with ipilimumab (ipi).
Groups:
- Phase 2, 8 mg Tilso/Ipi: IMO-2125 (tilso) intratumoral injection plus ipilimumab (ipi)
  IMO-2125 (tilso): Drug: IMO-2125 (tilso) (8 mg as the RP2D) Intratumoral injection administered as 9 doses on Weeks 1, 2, 3, 5, 8, 11, 17, 23, and 29.
  Ipilimumab (ipi): 4 doses administered intravenously at a dose of 3 mg/kg over 90 minutes on Weeks 2, 5, 8, and 11.
Period: Overall Study
Arm/Group | Phase 2, 8 mg Tilso/Ipi
Started | 53 (All participants who received at least 1 dose of study treatment (8 mg Tilso/Ipi) including nine rollover participants from the Phase 1 study.)
Completed | 18
Not Completed | 35
Not completed — Death | 26
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 2
Not completed — Protocol Violation | 1
Not completed — Progressive Disease | 1
Not completed — Study Terminated by Sponsor | 4

BASELINE CHARACTERISTICS:
Population: Includes all participants who received at least 1 dose of study treatment.
Groups:
- Phase 2, 8 mg Tilso/Ipi: IMO-2125 intratumoral injection plus ipilimumab
  IMO-2125: Drug: IMO-2125 (8 mg as the RP2D) Intratumoral injection administered as 9 doses on Weeks 1, 2, 3, 5, 8, 11, 17, 23, and 29.
  Ipilimumab: 4 doses administered intravenously at a dose of 3 mg/kg over 90 minutes on Weeks 2, 5, 8, and 11.
Arm/Group | Phase 2, 8 mg Tilso/Ipi
Number analyzed (Participants) | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.6 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 45
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 47
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 53
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Population: Not done for four participants.
  kg/m^2
    number analyzed (Participants) | 49
    (all) | 28.9 (6.4)
Baseline Melanoma Characteristics [Count of Participants; unit: Participants]
  Primary Histology - Cutaneous | 42
  Primary Histology - Mucosal | 5
  Primary Histology - Other | 6
Baseline Melanoma Stage [Count of Participants; unit: Participants] — Physician assessed and determined based on American Joint Committee on Cancer (AJCC) Staging System for Melanoma, Seventh Edition, which determines the stage (I-V) based on the TNM classification. T refers to tumor size, N refers to nearby lymph nodes and M represents metastasized (spread) to other parts of the body. This staging number is obtained as a sum of the TNM classification. The lower the number, the lower the cancer stage and the better the prognosis for the patient. The higher the stage, the worse the prognosis for the patient.
  Participants
    IIIA | 2
    IIIB | 2
    IIIC | 13
    IVM1A | 7
    IVM1B | 6
    IVM1C | 22
    Other: IV | 1
Baseline Brain Metastases [Count of Participants; unit: Participants]
  Yes | 2
  No | 49
  Unknown | 2
Baseline Visceral Metastases [Count of Participants; unit: Participants]
  Yes | 26
  No | 23
  Unknown | 4
Baseline Elevated LDH [Count of Participants; unit: Participants]
  Yes | 14
  No | 37
  Unknown | 2
Baseline BRAF Mutation [Count of Participants; unit: Participants]
  Yes | 23
  No | 26
  Unknown | 4
Prior Melanoma Treatment [Number; unit: prior treatments] — Indicates multiple, known prior melanoma treatments. Participants may be counted in more than one category based on combination of prior melanoma treatments.
  prior treatments
    Therapeutic Lymph Node Dissection | 23
    Radiation | 14
    Chemotherapy | 9
    Interferon | 9
    BRAF Inhibitor | 9
    MEK Inhibitor | 8
    CTLA-4 Inhibitor | 17
    PD-(L)1 Inhibitor | 49
    Other | 23

OUTCOME MEASURES:

1. Primary Outcome: Phase 2: Number of Participants With Objective Response Rate (ORR) Using RECIST v1.1
Description: The following combined analysis populations were used for outcome measures (efficacy analysis N=53):
  * The Phase 2, 8 mg Tilso/Ipi efficacy evaluable population (N=44)
  * The Phase 1, 8 mg Tilso/Ipi evaluable population (N=9)
  The ORR for 49 evaluable (4 non-evaluable) participants who received the recommended Phase 2 dose (RP2D) of 8 mg Tilso/Ipi was calculated using the participant's best overall response (BOR).
  Per Response Evaluation Criteria in Solid Tumors (RECIST v1.1) for target lesions as assessed by MRI, CT or X-ray: Complete Response (CR) - disappearance of all target lesions; Partial Response (PR) - >=30% decrease from baseline of the sum of diameters of all target lesions; Stable Disease (SD) - does not qualify for CR, PR or Progression; Progressive Disease (PD) - 20% increase in the sum of diameters of target lesions.
  Overall Response = CR or PR
Time Frame: 33 weeks (29 weeks of treatment, 4 weeks follow up)
Population: Per the SAP, section 6, Analysis Populations used for efficacy, the analysis populations utilize both PIIEE (Primary Ipilimumab + IMO-2125 Efficacy Evaluable) who are ipilimumab-naive and SIIEE (Secondary Ipilumumab + IMO-2125 Efficacy Evaluable) who are not ipilumumab-naive that were treated at the RP2D, regardless of phase, and received at least one dose of each study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 2, 8 mg Tilso/Ipi: Arm/Group includes 9 participants rolled over from Phase 1 8mg Tilso/Ipi
  IMO-2125 (tilso) intratumoral injection plus ipilimumab (ipi)
  IMO-2125 (tilso): Drug: IMO-2125 (tilso) (8 mg as the RP2D) Intratumoral injection administered as 9 doses on Weeks 1, 2, 3, 5, 8, 11, 17, 23, and 29.
  Ipilimumab (ipi): 4 doses administered intravenously at a dose of 3 mg/kg over 90 minutes on Weeks 2, 5, 8, and 11.
Arm/Group | Phase 2, 8 mg Tilso/Ipi
Number analyzed (Participants) | 53
Participants
  Complete Response | 2
  Partial Response | 9
  Stable Disease | 24
  Progressive Disease | 14
  Non-evaluable | 4
Statistical Analysis 1: Comparison: Phase 2, 8 mg Tilso/Ipi; Testing the best overall confirmed response rate against the historical control rate of 0.11 (extracted from the literature review); Test type: Other — Estimation; p = 0.0158, One-sided Clopper-Pearson test — P-value of the overall response tested against the null rate of 11% based on 1-sided exact (Clopper-Pearson) test

2. Secondary Outcome: Phase 2: Progression-free Survival
Description: The following combined analysis populations were used for outcome measures (efficacy analysis N=53):
  * The Phase 2, 8 mg Tilso/Ipi efficacy evaluable population N=40 (44 with 4 non-evaluable)
  * The Phase 1, 8 mg Tilso/Ipi evaluable population (N=9)
  Progression-free survival was defined as the number of months from the initiation of treatment to confirmed disease progression using RECIST v1.1 or death from any cause.
Time Frame: 33 weeks (29 weeks of treatment, 4 weeks follow up)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2, 8 mg Tilso/Ipi
Number analyzed (Participants) | 53
Participants
  Participants with disease progression or death | 41
  Participants who did not progress or die | 8
  Non-evaluable | 4
Statistical Analysis 1: Comparison: Phase 2, 8 mg Tilso/Ipi; Test type: Other — Estimation; Kaplan-Meier = 5.06, 95% CI 2-sided [3.65 to 7.00] — Kaplan-Meier estimate of median PFS in months

3. Secondary Outcome: Phase 2: Overall Survival - 6 Months
Description: The following combined analysis populations were used for outcome measures (efficacy analysis N=53):
  * The Phase 2, 8 mg Tilso/Ipi efficacy evaluable population N=44 (40 with 4 non-evaluable)
  * The Phase 1, 8 mg Tilso/Ipi evaluable population (N=9)
  Overall survival was defined as the number of months from initiation of treatment to death from any cause.
Time Frame: 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2, 8 mg Tilso/Ipi
Number analyzed (Participants) | 53
Participants
  Participants who died at or before 6 months | 6
  Participants who did not die at or before 6 months | 43
  Non-evaluable | 4
Statistical Analysis 1: Comparison: Phase 2, 8 mg Tilso/Ipi; Test type: Other — Landmark analysis of overall survival at six (6) months; Kaplan-Meier = 87.5, 95% CI 2-sided [74.3 to 94.2] — Kaplan-Meier estimate of percentage of participants surviving at six (6) months

4. Secondary Outcome: Phase 2: Overall Survival - 12 Months
Description: The following combined analysis populations were used for outcome measures (efficacy analysis N=53):
  * The Phase 2, 8 mg Tilso/Ipi efficacy evaluable population N=40 (44 with 4 non-evaluable)
  * The Phase 1, 8 mg Tilso/Ipi evaluable population (N=9)
  Overall survival was defined as the number of months from initiation of treatment to death from any cause.
Time Frame: 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2, 8 mg Tilso/Ipi
Number analyzed (Participants) | 53
Participants
  Participants who died at or before 12 months | 19
  Participants who did not die at or before 12 months | 30
  Non-evaluable | 4
Statistical Analysis 1: Comparison: Phase 2, 8 mg Tilso/Ipi; Test type: Other — Landmark analysis of overall survival at twelve (12) months; Kaplan-Meier = 60.0, 95% CI 2-sided [44.7 to 72.4] — Kaplan-Meier estimate of percentage of participants surviving at twelve (12) months

ADVERSE EVENTS:
Time Frame: From the signing of informed consent to the end of the study (up to 12 months), which entails up to 29 weeks of treatment, a safety follow-up visit at week 32 and ongoing follow-up every 3 months until documented disease progression, new melanoma treatment, withdrawal of consent or death.
Description: Definitions aligned with FDA and ICH requirements.
Groups:
- Phase 2, 8 mg Tilso/Ipi: Arm/Group includes 9 participants rolled over from Phase 1, 8 mg Tilso/Ipi.
  IMO-2125 intratumoral injection plus ipilimumab
  IMO-2125: Drug: IMO-2125 (8 mg as the RP2D) Intratumoral injection administered as 9 doses on Weeks 1, 2, 3, 5, 8, 11, 17, 23, and 29.
  Ipilimumab: 4 doses administered intravenously at a dose of 3 mg/kg over 90 minutes on Weeks 2, 5, 8, and 11.
Arm/Group | Phase 2, 8 mg Tilso/Ipi
All-Cause Mortality (participants affected / at risk) | 26/53
Serious Adverse Events (participants affected / at risk) | 15/53
Other Adverse Events (participants affected / at risk) | 52/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 2, 8 mg Tilso/Ipi (N=53)
Hyponatraemia (Metabolism and nutrition disorders) | 1
Urinary tract infection (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Anaphylactic reaction (Immune system disorders) | 1
Asthenia (General disorders) | 1
Autoimmune colitis (Gastrointestinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Depressed level of consciousness (Nervous system disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Influenza like illness (General disorders) | 1
Large intestine perforation (Gastrointestinal disorders) | 1
Skin neoplasm bleeding (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hypophysitis (Endocrine disorders) | 1
Abdominal mass (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastritis haemorrhagic (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 1
Autoimmune hepatitis (Hepatobiliary disorders) | 1
Clostridium difficile infection (Infections and infestations) | 1
Pleural infection (Infections and infestations) | 1
Failure to thrive (Metabolism and nutrition disorders) | 1
Guillain-Barre syndrome (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 2, 8 mg Tilso/Ipi (N=53)
Fatigue (General disorders) | 30
Pyrexia (General disorders) | 18
Chills (General disorders) | 15
Influenza like illness (General disorders) | 10
Injecion site pain (General disorders) | 5
Injection site reaction (General disorders) | 4
Pain (General disorders) | 3
Alanine aminotransferase increased (Investigations) | 16
White blood cell count decreased (Investigations) | 13
Aspartate aminotransferase increased (Investigations) | 13
Lymphocyte count decreased (Investigations) | 13
Blood creatinine increased (Investigations) | 9
Gamma-glutamyltransferase increased (Investigations) | 9
Platelet count decreased (Investigations) | 6
Blood alkaline phosphatase increased (Investigations) | 5
Neutrophil count decreased (Investigations) | 4
Decreased appetite (Metabolism and nutrition disorders) | 13
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 9
Hypophosphataemia (Metabolism and nutrition disorders) | 7
Hyponatraemia (Metabolism and nutrition disorders) | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 7
Hyperkalaemia (Metabolism and nutrition disorders) | 5
Hypoalbumanaemia (Metabolism and nutrition disorders) | 6
Hypokalaemia (Metabolism and nutrition disorders) | 6
Dehydration (Metabolism and nutrition disorders) | 4
Hyperuricaemia (Metabolism and nutrition disorders) | 3
Nausea (Gastrointestinal disorders) | 22
Diarrhoea (Gastrointestinal disorders) | 22
Vomiting (Gastrointestinal disorders) | 15
Constipation (Gastrointestinal disorders) | 6
Abdominal pain (Gastrointestinal disorders) | 3
Colitis (Gastrointestinal disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 15
Pruritus (Skin and subcutaneous tissue disorders) | 11
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3
Anaemia (Blood and lymphatic system disorders) | 19
Headache (Nervous system disorders) | 16
Dizziness (Nervous system disorders) | 9
Paraesthesia (Nervous system disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Urinary tract infection (Infections and infestations) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5
Flushing (Vascular disorders) | 3
Hypophysitis (Endocrine disorders) | 4
Depression (Psychiatric disorders) | 4
Anxiety (Psychiatric disorders) | 3

LIMITATIONS AND CAVEATS:
The analysis populations, as defined in section 6 of the Statistical Analysis Plan, analyzed participants enrolled in the phase 2 study (N=44) and participants rolled in from the phase 1, 8 mg Tilso/Ipi population (N=9).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-03-27): https://cdn.clinicaltrials.gov/large-docs/67/NCT02644967/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-05): https://cdn.clinicaltrials.gov/large-docs/67/NCT02644967/SAP_001.pdf